CLINICAL TRIAL: NCT04855266
Title: A Randomized, Controlled, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy of Intravenous Iron Sucrose in Patients With Non-anemic Iron Deficiency and Postural Orthostatic Tachycardia Syndrome (POTS)
Brief Title: Iron Sucrose in Patients With Iron Deficiency and POTS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kamal Shouman, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-000488
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Iron-deficiency; Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Anemia, Iron-Deficiency; Postural Orthostatic Tachycardia Syndrome | interventions — Sucrose; Ferric Oxide, Saccharated; Tilt-Table Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron Sucrose Group (Experimental): Subjects will receive intravenous iron sucrose during a tilt table test
  Interventions: Drug: Sucrose; Diagnostic Test: Tilt Table Test
- Placebo Group (Placebo Comparator): Subjects will receive intravenous placebo during a tilt table test
  Interventions: Drug: Placebo; Diagnostic Test: Tilt Table Test

INTERVENTIONS:
Drug: Sucrose — 5 mg/kg of intravenous iron sucrose (maximum dose of 200 mg). Iron sucrose will be diluted
  Other Names: Venofer
  Arms: Iron Sucrose Group
Drug: Placebo — Normal saline (NaCl 0.9%) 5 mL/kg (maximum volume 210 mL)
  Arms: Placebo Group
Diagnostic Test: Tilt Table Test — A table that adjusts the body position from horizontal to vertical to simulate standing up. Heart rate and blood pressure are monitored throughout the test.

SUMMARY:
This study aims to investigate whether the treatment of non-anemic iron deficiency with intravenous iron sucrose will result in decreased symptom reporting and improved cardiovascular indices in patients with Postural Orthostatic Tachycardia syndrome (POTS).

ELIGIBILITY:
Inclusion Criteria:

* Patients (age 12 to years and older) with chronic (>3 months) symptoms of orthostatic intolerance, including but not limited to lightheadedness, syncope, headache, fatigue, weakness, sweating, nausea and heart palpitations.
* Symptomatic orthostatic heart rate increment ≥30 bpm if >19 years old or ≥40 bpm if <19 years old during a 10 minute 70 degree head up tilt study
* Presence of non-anemic iron deficiency, defined as serum ferritin levels <20 ug/L with hemoglobin no less than 1 gm/dL below the normal reference range as defined for age and gender
* Consent obtained from responsible guardian AND from subjects, 12-17 years of age
* Consent obtained for subjects 18 years of age and older

Exclusion Criteria:

* Orthostatic hypotension (decrease of systolic BP>30 mmHg and/or diastolic BP>15mmHg within 3 minutes of 70 degree head up tilt study)
* Pregnant or lactating females
* The presence of failure of other organ systems or systemic illness that can affect autonomic function
* Concomitant therapy with anticholinergic, alpha-adrenergic antagonists, beta-adrenergic antagonists or other medications which could interfere with autonomic testing. Patients may participate if the potentially interfering medication is held for five half-lives prior to the study
* Laboratory evidence of anemia or iron overload
* Personal history of hematochromatosis or first degree relative with hematochromatosis
* Known sensitivity to Venofer® (iron sucrose injection, USP) or other intravenous iron preparation

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change in autonomic dysfunction symptoms | Baseline, 7 days, 6 months
  Measured using the self-reported Composite Autonomic Symptom Score (COMPASS) questionnaire that asks 31 questions regarding symptoms of autonomic dysfunction
Change in postural heart rate increase | Baseline, 7 days
  Heart rate change during tilt table test measured in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Shouman, MD, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials